CLINICAL TRIAL: NCT00088023
Title: A Phase I Study of PT-523 in Patients With Solid Tumors
Brief Title: Safety Study of PT-523 in Cancer Patients to Treat Solid Tumors Including a Preliminary Assessment of Effectiveness
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-000; DFCI Legacy- 03-183; CTEP Grant No.- UO1-CA62490-09; NSC No.- 712783
Record Dates: First submitted 2004-07-19; First posted 2004-07-20 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Neoplasms
Keywords: Solid tumors
MeSH Terms: conditions — Neoplasms | interventions — N(alpha)-(4-amino-4-deoxypteroyl)-N(delta)-hemiphthaloyl-L-ornithine; Injections

INTERVENTIONS:
Drug: PT-523 for Injection

SUMMARY:
The purpose of this study is to determine the safety of a short intravenous infusion of PT-523 to patients with solid tumors who have failed curative or survival prolonging therapy or for whom no such therapies exist.

DETAILED DESCRIPTION:
The primary objectives of this study are 1) to evaluate the safety of a short intravenous infusion of PT-523 when administered on days 1, 8, and 15 of a 28-day cycle to patients with solid tumors who have failed curative or survival prolonging therapy or for whom no such therapies exist; and 2) to establish the maximum tolerated dose (MTD) and identify the dose limiting toxicities (DLT) of PT-523.

The secondary objectives of this study are to determine the pharmacokinetics and to evaluate preliminary efficacy of PT-523.

ELIGIBILITY:
Inclusion Criteria:

* Presence of metastatic or inoperable malignancy, other than leukemia or a primary central nervous system (CNS) tumor, for which there is no known curative or survival prolonging palliative therapy, or failure of these therapies .
* Age greater than or equal to 18 years.
* Life expectancy greater than or equal to 2 months.
* ECOG performance status 0 - 2.
* Adequate organ function and bone marrow reserve.
* Use of appropriate contraceptive method.
* Sign patient informed consent.

Exclusion Criteria:

* Active brain metastases.
* Presence of third-space fluid collections (pleural effusion, ascites).
* Major surgery within 3 weeks prior to dosing.
* Prior chemotherapy or radiation therapy within 3 weeks prior to dosing (6 weeks for nitrosoureas or mitomycin-C). Prior antifolate therapy is permitted, as long as it has not been administered within 3 weeks prior to dosing with PT-523.
* Prior bone marrow transplantation.
* Presence of uncontrolled serious medical or psychiatric illness.
* Patients requiring radiation therapy.

There are no limitations on the extent or type of prior therapy received by the patient other than the time intervals indicated above, as long as the patient has demonstrated complete recovery from any adverse effects, and fulfills all relevant inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-03; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Paul Eder, M.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- See also: Hana Biosciences, Inc. is a South San Francisco, CA-based biopharmaceutical company that acquires, develops, and commercializes innovative products to advance cancer care. — http://www.hanabiosciences.com